CLINICAL TRIAL: NCT01713231
Title: Effect of High-Dose Vitamin D on Bone Density in Osteogenesis Imperfecta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louis-Nicolas Veilleux Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Louis-Nicolas Veilleux Ph.D., postdoctoral fellow, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A02-M14-12A
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: osteogenesis imperfecta; high-dose vitamin D; bone density; muscle function
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard-dose vitamin D (Active Comparator): one group of 30 participants will be randomized to receive vitamin D3 at a dose of 400 international units per day ('standard-dose group').
  Interventions: Dietary Supplement: standard-dose vitamin D (400IU per day)
- high-dose vitamin D (Experimental): One group of 30 participants will be randomized to receive vitamin D3 at a dose of 2000 international units per day ('high-dose group').
  Interventions: Dietary Supplement: high-dose vitamin D (2000 IU per day)

INTERVENTIONS:
Dietary Supplement: standard-dose vitamin D (400IU per day)
  Arms: standard-dose vitamin D
Dietary Supplement: high-dose vitamin D (2000 IU per day)
  Arms: high-dose vitamin D

SUMMARY:
* Overall Objective: To test the hypothesis that oral vitamin D supplementation at higher than currently prescribed doses has a beneficial effect on the skeleton of young patients with osteogenesis imperfecta (OI).
* Specific Aims: 1. To determine whether 12 months of high-dose vitamin D supplementation, compared to standard-dose vitamin D supplementation, increases areal bone mineral density z-scores at the lumbar spine. 2. To examine the effectiveness of high-dose vitamin D supplementation to increase trabecular and cortical bone mineral density at the radius. 3. To examine whether high-dose vitamin D supplementation has an effect on physiological determinants of bone mass (parathyroid hormone, activity of bone metabolism, muscle function).
* Background: In a preliminary cross-sectional study of 282 OI patients we observed an inverse relationship between serum 25-hydroxyvitamin D and parathyroid hormone levels and a positive relationship between circulating levels of 25-hydroxyvitamin D and lumbar spine areal bone mineral density z-scores. This suggested that high-dose vitamin D supplementation would have a beneficial effect on bone density. Most OI patients currently receive oral vitamin D supplementation of 400 International Units per day, but doses of 2000 International Units per day are safe and have been shown to be beneficial in studies on healthy adolescents.
* Study Design: This is a parallel-group double-blind randomized controlled trial of 12 months duration on 60 children and adolescents aged 6 to 19 years with a clinical diagnosis of OI. One group of 30 participants will be randomized to receive vitamin D3 at a dose of 2000 international units per day ('high-dose group'). The other group of 30 participants will be randomized to receive vitamin D3 at a dose of 400 international units per day ('standard-dose group'). Randomization will be stratified according to pubertal status and bisphosphonate treatment status.
* Clinical Relevance: The proposed study aims at direct improvements in the care of OI patients. If a simple and low-cost 'intervention' such as high-dose vitamin D supplementation can be shown to be effective in relieving some of the disease burden associated with OI, the benefit to OI patients worldwide would be substantial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OI of any type.

Exclusion Criteria:

* Any condition that renders bone density measurements at the lumbar spine impossible. An example for this is prior spinal fusion surgery.
* Bisphosphonate therapy for less than two years duration.
* Use of medication, other than bisphosphonates, known to affect bone metabolism or 25OHD serum concentrations. Examples are anti-epileptics, active vitamin D metabolites, corticosteroids and thyroid hormones.
* Liver and renal disease known to interfere with vitamin D metabolism.
* Any other disorder of calcium and phosphate metabolism (apart from vitamin D deficiency) that might interfere with PTH.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in areal bone mineral density z-score of the lumbar spine | at baseline and 12 months
  LS-aBMD z-score will be used as the primary outcome.The lumbar spine is the standard site of measurement both in the clinical follow up of OI patients .

SECONDARY OUTCOMES:
Change in trabecular and cortical volumetric bone mineral density z-scores at the radius, as measured by pQCT, relative to baseline. | at baseline and at 12 months
  Trabecular bone is analyzed at the distal radial metaphysis ('4% site'). Cortical bone is analyzed at the radial diaphysis ('65% site').

OTHER OUTCOMES:
Percentage change in lower extremity muscle power per body weight, as measured by jumping mechanography, relative to baseline. | baseline and 12 months
  A countermovement jump to maximal height ('single two-legged jump') will be evaluated. In patients who are unable to jump, the heel-rise test will be used to determine muscle power.

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospitals for Children-Canada, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Plante L, Veilleux LN, Glorieux FH, Weiler H, Rauch F. Effect of high-dose vitamin D supplementation on bone density in youth with osteogenesis imperfecta: A randomized controlled trial. Bone. 2016 May;86:36-42. doi: 10.1016/j.bone.2016.02.013. Epub 2016 Feb 24. PMID 26924265